CLINICAL TRIAL: NCT02107443
Title: Improving Communication for Cancer Treatment: Addressing Concerns of Older Cancer Patients and Caregivers
Brief Title: Improving Communication in Older Cancer Patients and Their Caregivers
Acronym: COACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Supriya Mohile (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor-Investigator, Supriya Mohile, Professor, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: URCC13070; NCI-2014-00619 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); URCC 13070 (Other: University of Rochester); URCC-13070 (Other: DCP); URCC-13070 (Other: CTEP); UG1CA189961 (NIH); U10CA037420 (NIH); CD-12-11-4634 (Other: PCORI)
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Adult Solid Neoplasm; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Geriatric Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I: Geriatric Assessment Intervention (Experimental): At the first study visit with their oncologist, patients and their caregivers (if participating) complete the GA and receive the intervention; GA summary plus GA targeted recommendations which is provided to the oncology team to discuss and implement if they so choose.
  Interventions: Behavioral: Geriatric Assessment Summary; Behavioral: Geriatric Assessment Targeted Recommendations; Behavioral: Geriatric Assessment (GA)
- Arm II: Usual Care (Active Comparator): At the first study visit with their oncologist, patients and their caregivers (if participating) complete the GA (no GA summary or recommendations are provided).
  Interventions: Behavioral: Geriatric Assessment (GA)

INTERVENTIONS:
Behavioral: Geriatric Assessment Summary — Complete summary of results from the Geriatric Assessment
  Arms: Arm I: Geriatric Assessment Intervention
Behavioral: Geriatric Assessment Targeted Recommendations — Recommendations are made based on areas patients were impaired in on the Geriatric Assessment. They include referrals, tests, medication review, instructions, and support services. The choice of which recommendation to implement is left to the discretion of the physician.
  Treatment modifications
  Arms: Arm I: Geriatric Assessment Intervention
Behavioral: Geriatric Assessment (GA) — A GA measures the issues important to older patients, including function, psychological status, cognitive abilities, social support, and the impact of medical problems on quality of life.

SUMMARY:
Over 60% of cancers occur in older persons, and the number of older persons with cancer is expected to grow as the population ages. Oncology clinical trials have traditionally excluded older patients with advanced cancer and chronic health conditions. In this context, where data is limited and risk from treatment is high, older patients with advanced cancer and their caregivers must understand how cancer treatment can affect quality of life in light of underlying health status. Better communication about age-related health conditions between oncologists, older patients with advanced cancer, and their caregivers may improve decision-making for cancer treatment and quality of life. A geriatric assessment (GA), a validated set of patient-centered outcomes, has been shown to identify concerns (e.g., function, cognition) important to older persons with cancer and their caregivers. In this cluster randomized clinical trial we examined whether providing a web-generated GA summary with targeted recommendations to older patients with advanced cancer, their caregivers, and their oncologists can improve communication about age-related concerns that could affect efficacy and tolerance of cancer treatment. We also determined whether the intervention improves patient-reported quality of life and patient and caregiver satisfaction.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Primary Aim - Direct Communication about Age-related Concerns: To determine if providing GA summary plus GA-driven recommendations to patients, their caregivers, and oncology physicians increases discussions about age-related issues during clinic consultation. [Patient-Centered Outcomes Research Institute (PCORI) specified]

II. Primary Aim - Patient Satisfaction with Communication about Age-related Concerns: To determine if providing geriatric assessment (GA) summary plus GA-driven recommendations to patients, their caregivers and oncology physicians improves patient satisfaction with communication with the oncology physician regarding age-related concerns. [National Cancer Institute (NCI) specified]

III. Secondary Aim - To determine whether initially providing patients, their caregivers, and oncology physicians with GA summary plus GA-driven recommendations prior to their treatment influences quality of life of older patients receiving treatment and their caregivers.

IV. Secondary Aim - To determine whether providing patients, their caregivers, and oncology physicians with GA summary plus GA-driven recommendations influences caregiver satisfaction with communication about age-related issues.

OUTLINE: Patients are randomized to 1 of 2 arms.

Arm I: At the first study visit with their oncologist, patients and their caregivers (if participating) complete the GA and receive the GA summary plus GA targeted recommendations which is provided to the oncology team to discuss and implement if they so choose.

Arm II: At the first study visit with their oncologist, patients and their caregivers (if participating) complete the GA (no GA summary or recommendations are provided).

Patients are followed at 4-6 weeks, 3 months, and 6 months. Survival data will be collected at 1 year after enrollment.

ELIGIBILITY:
Inclusion Criteria for Patients

* Male or female 70 years of age or older
* Diagnosis of an advanced solid tumor malignancy (advanced cancer) or lymphoma. In most situations, this would be a stage IV cancer. A patient with a diagnosis of stage III cancer or lymphoma is eligible if cure is not possible or anticipated. Clinical staging without pathological confirmation of advanced disease is allowed.
* Must be considering or currently receiving any kind of cancer treatment (any line), including but not limited to hormonal treatment, chemotherapy, monoclonal antibody therapy, or targeted therapy. Patients who are considering therapy are eligible even if they ultimately choose not to be on therapy. Patients with a history of any previous cancer treatment, including radiation and/or surgery are eligible. A patient may also be enrolled on a treatment trial and participate in this study, if all other inclusion and exclusion criteria are met.
* Have at least one geriatric assessment domain meet the cut-off score for impairment other than polypharmacy.
* Have visits planned with the oncology physician for at least 3 months and be willing to come in for study visits.
* Able to provide informed consent or, if the oncology physician determines the patient to not have decision-making capacity, a patient-designated health care proxy (per institutional policies) must sign consent by the baseline visit.
* Subject has adequate understanding of the English language because not all GA measures have been validated in other languages.

Exclusion Criteria for Patients

* Have surgery planned within 3 months of consent. Patients who have previously received surgery are eligible.
* Have already made a decision to not undergo any cancer treatment (e.g., being followed in best supportive care or hospice).

Inclusion Criteria for Caregivers

* Selected by the patient when asked if there is a "family member, partner, friend or caregiver [age 21 or older] with whom you discuss or who can be helpful in health-related matters;" patients who cannot identify such a person ("caregiver") can be eligible for the study. A caregiver need not be someone who lives with the patient or provides direct hands-on care. A caregiver can be any person who provides support (in any way) to the patient.
* If a health care proxy signs consent for or with a patient, and wants to participate in the caregiver portion of the study, this same person will always be the caregiver selected. If a health care proxy does not want to enroll as a caregiver in the study or, if enrolled, chooses to stop their own participation in the caregiver portion of the study, but is able to assist the patient in completing the study, the patient can still participate. In other words, the health care proxy can choose NOT to participate in the caregiver portion of the study. This does not preclude the patient from participating in the patient portion of the study with the health care proxy's assistance.

Exclusion Criteria for Caregivers

-Caregivers unable to understand the consent form due to cognitive, health, or sensory impairment will be excluded.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 546 (Actual)
Dates: Start 2014-10-27 (Actual); Primary Completion 2017-05-12 (Actual); Study Completion 2020-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Supriya Mohile, Principal Investigator — University of Rochester NCORP Research Base
Locations (19):
- United States (19):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Delaware/Christiana Care NCORP, Newark, Delaware
  - Hawaii, Honolulu, Hawaii
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Heartland NCORP, Decatur, Illinois
  - Kansas City NCORP, Prairie Village, Kansas
  - Wichita NCORP, Wichita, Kansas
  - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Metro-Minnesota NCORP, Minneapolis, Minnesota
  - Nevada NCORP, Las Vegas, Nevada
  - Northwell Health, Lake Success, New York
  - University of Rochester, Rochester, New York
  - Southeast Clinical Oncology Research Consortium, Winston-Salem, North Carolina
  - Columbus NCORP, Columbus, Ohio
  - Pacific Cancer Research Consortium Ncorp, Portland, Oregon
  - Geisinger Cancer Institute NCORP, Danville, Pennsylvania
  - Greenville NCORP, Greenville, South Carolina
  - WiNCORP, Marshfield, Wisconsin
  - Aurora NCORP, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Kehoe LA, Sohn MB, Wang L, Mohile S, Kamen C, Van Orden K, Wells M, Gilmore N, Arana-Chicas E, Gudina A, Yilmez S, Griggs L, Loh KP. Associations of quality of social support and accurate beliefs about curability among older adults with advanced cancer. J Geriatr Oncol. 2024 Nov;15(8):102061. doi: 10.1016/j.jgo.2024.102061. Epub 2024 Sep 10. PMID 39260086
- [Derived] Singhal S, Wang Y, Qin Z, Peterson DR, Dunne RF, Culakova E, Hopkins JO, Melnyk N, Onitilo A, Targia V, Mohile S, Loh KP. Nutritional impairment, psychological health and quality of life among older adults with advanced cancer: A secondary analysis of a randomized clinical trial. Cancer Med. 2024 Jun;13(12):e7348. doi: 10.1002/cam4.7348. PMID 38898664
- [Derived] Lund JL, Cacciatore J, Tylock R, Su IH, Sharma S, Hinton SP, Smith S, Nowels MA, Chen X, Duberstein PR, Hanson LC, Mohile SG. Development and Evaluation of a Multisource Approach to Extend Mortality Follow-Up for Older Adults With Advanced Cancer Enrolled in Randomized Trials. JCO Clin Cancer Inform. 2024 Apr;8:e2300183. doi: 10.1200/CCI.23.00183. PMID 38564692
- [Derived] Jensen-Battaglia M, Mohammed M, Loh KP, Wells M, Tylock R, Ramsdale E, Canin B, Geer J, O'Rourke MA, Liu JJ, Seplaki CL, Mohile SG, Wildes TM. Modifiable fall risk factors among older adults with advanced cancer: Secondary analysis of a cluster-randomized clinical trial. J Geriatr Oncol. 2023 Nov;14(8):101650. doi: 10.1016/j.jgo.2023.101650. Epub 2023 Oct 26. PMID 37897888
- [Derived] Jensen-Battaglia M, Lei L, Xu H, Loh KP, Wells M, Tylock R, Ramsdale E, Kleckner AS, Mustian KM, Dunne RF, Kehoe L, Bearden J 3rd, Burnette BL, Whitehead M, Mohile SG, Wildes TM. Communication About Fall Risk in Community Oncology Practice: The Role of Geriatric Assessment. JCO Oncol Pract. 2022 Oct;18(10):e1630-e1640. doi: 10.1200/OP.22.00173. Epub 2022 Aug 19. PMID 35984998
- [Derived] Jensen-Battaglia M, Lei L, Xu H, Kehoe L, Patil A, Loh KP, Ramsdale E, Magnuson A, Kleckner AS, Wildes TM, Lin PJ, Mustian KM, Giri G, Whitehead M, Bearden J 3rd, Burnette BL, Geer J, Mohile SG, Dunne RF. Association of Oncologist-Patient Communication With Functional Status and Physical Performance in Older Adults: A Secondary Analysis of a Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e223039. doi: 10.1001/jamanetworkopen.2022.3039. PMID 35302628
- [Derived] Loh KP, Seplaki CL, Sanapala C, Yousefi-Nooraie R, Lund JL, Epstein RM, Duberstein PR, Flannery M, Culakova E, Xu H, McHugh C, Klepin HD, Lin PJ, Watson E, Grossman VA, Liu JJ, Geer J, O'Rourke MA, Mustian K, Mohile SG. Association of Prognostic Understanding With Health Care Use Among Older Adults With Advanced Cancer: A Secondary Analysis of a Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 Feb 1;5(2):e220018. doi: 10.1001/jamanetworkopen.2022.0018. PMID 35179585
- [Derived] Gilmore N, Xu H, Kehoe L, Kleckner AS, Moorthi K, Lei L, Mohamed MRS, Loh KP, Culakova E, Flannery M, Ramsdale E, Duberstein PR, Canin B, Kamen C, Giri G, Watson E, Patil A, Onitilo AA, Burnette B, Janelsins M, Mohile SG. Evaluating the association of frailty with communication about aging-related concerns between older patients with advanced cancer and their oncologists. Cancer. 2022 Mar 1;128(5):1101-1109. doi: 10.1002/cncr.34010. Epub 2021 Nov 11. PMID 34762734
- [Derived] Flannery MA, Mohile S, Culakova E, Norton S, Kamen C, Dionne-Odom JN, DiGiovanni G, Griggs L, Bradley T, Hopkins JO, Liu JJ, Loh KP. Completion of Patient-Reported Outcome Questionnaires Among Older Adults with Advanced Cancer. J Pain Symptom Manage. 2022 Feb;63(2):301-310. doi: 10.1016/j.jpainsymman.2021.07.032. Epub 2021 Aug 8. PMID 34371137
- [Derived] Kleckner AS, Wells M, Kehoe LA, Gilmore NJ, Xu H, Magnuson A, Dunne RF, Jensen-Battaglia M, Mohamed MR, O'Rourke MA, Vogelzang NJ, Dib EG, Peppone LJ, Mohile SG. Using Geriatric Assessment to Guide Conversations Regarding Comorbidities Among Older Patients With Advanced Cancer. JCO Oncol Pract. 2022 Jan;18(1):e9-e19. doi: 10.1200/OP.21.00196. Epub 2021 Jul 6. PMID 34228510
- [Derived] Xu H, Kadambi S, Mohile SG, Yang S, Kehoe LA, Wells M, Culakova E, Kamen C, Obrecht S, Mohamed M, Gilmore NJ, Magnuson A, Grossman VA, Hopkins JO, Geer J, Berenberg J, Mustian K, Cupertino A, Mohile N, Loh KP. Caregiving burden of informal caregivers of older adults with advanced cancer: The effects of rurality and education. J Geriatr Oncol. 2021 Sep;12(7):1015-1021. doi: 10.1016/j.jgo.2021.04.002. Epub 2021 Apr 12. PMID 33858803
- [Derived] Mohile SG, Epstein RM, Hurria A, Heckler CE, Canin B, Culakova E, Duberstein P, Gilmore N, Xu H, Plumb S, Wells M, Lowenstein LM, Flannery MA, Janelsins M, Magnuson A, Loh KP, Kleckner AS, Mustian KM, Hopkins JO, Liu JJ, Geer J, Gorawara-Bhat R, Morrow GR, Dale W. Communication With Older Patients With Cancer Using Geriatric Assessment: A Cluster-Randomized Clinical Trial From the National Cancer Institute Community Oncology Research Program. JAMA Oncol. 2020 Feb 1;6(2):196-204. doi: 10.1001/jamaoncol.2019.4728. PMID 31697365
- [Derived] Kehoe LA, Xu H, Duberstein P, Loh KP, Culakova E, Canin B, Hurria A, Dale W, Wells M, Gilmore N, Kleckner AS, Lund J, Kamen C, Flannery M, Hoerger M, Hopkins JO, Liu JJ, Geer J, Epstein R, Mohile SG. Quality of Life of Caregivers of Older Patients with Advanced Cancer. J Am Geriatr Soc. 2019 May;67(5):969-977. doi: 10.1111/jgs.15862. Epub 2019 Mar 29. PMID 30924548
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (GA Informational Intervention): Patients and their caregivers (if participating) complete the GA and receive the GA summary and recommendations guided by GA results provided by the oncology team to discuss and implement for each age-related issue at baseline.
  Informational Intervention: Complete GA summary plus GA-driven recommendations
- Arm II (Usual Care): Patients and their caregivers (if participating) complete the GA at baseline.
Period: Overall Study
Arm/Group | Arm I (GA Informational Intervention) | Arm II (Usual Care)
Started | 296 | 250
Completed | 198 | 167
Not Completed | 98 | 83
Not completed — Death | 42 | 30
Not completed — Study Protocol Violation | 3 | 1
Not completed — Registered but Not Eligible | 0 | 1
Not completed — Withdrawal: Hospitalization/Hospice | 28 | 28
Not completed — Withdrawal: Disliked Study Procedures | 1 | 2
Not completed — Withdrawal: Changed Mind | 2 | 0
Not completed — Withdrawal: Changed MD/Facility | 1 | 3
Not completed — Withdrawal: Too Many Forms | 3 | 1
Not completed — Withdrawal: Too Time Consuming | 3 | 6
Not completed — Withdrawal: Feeling Overwhelmed | 2 | 1
Not completed — Withdrawal: Other Medical | 9 | 5
Not completed — Withdrawal: Disease Progression | 4 | 2
Not completed — Withdrawal: Personal Issues | 0 | 3

BASELINE CHARACTERISTICS:
Population: * Non-Evaluable Patients: Arm I- 3 Patients Study Protocol Violation; Arm II- 1 Patient Study Protocol Violation, 1 Patient Registered then found to be ineligible.
  * Missing Demographics information from 1 evaluable patient from Arm I. This is denoted as Unknown.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (GA Informational Intervention) | Arm II (Usual Care) | Total
Number analyzed (Participants) | 293 | 248 | 541
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One subject did not provide demographic information in Arm I.
  years
    number analyzed (Participants) | 292 | 248 | 540
    (all) | 76.71 (5.19) | 76.41 (5.27) | 76.57 (5.22)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 137 | 127 | 264
  Gender: Male | 155 | 121 | 276
  Gender: Unknown | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic White | 263 | 219 | 482
  Race/Ethnicity: African American | 19 | 21 | 40
  Race/Ethnicity: Other | 10 | 8 | 18
  Race/Ethnicity: Unknown | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 293 | 248 | 541
Marital Status [Count of Participants; unit: Participants]
  Single, Never Married | 3 | 4 | 7
  Married | 192 | 148 | 340
  Separated | 1 | 7 | 8
  Domestic Partnership | 2 | 6 | 8
  Widowed | 59 | 50 | 109
  Divorced | 35 | 33 | 68
  Unknown | 1 | 0 | 1
Education [Count of Participants; unit: Participants]
  Less than High School | 36 | 30 | 66
  High School | 114 | 81 | 195
  More than High School | 142 | 137 | 279
  Unknown | 1 | 0 | 1
Cancer Type [Count of Participants; unit: Participants]
  Breast | 31 | 38 | 69
  Gastrointestinal | 72 | 66 | 138
  Genitourinary | 46 | 33 | 79
  Gynecological | 22 | 12 | 34
  Lung | 78 | 62 | 140
  Lymphoma | 23 | 18 | 41
  Other | 20 | 19 | 39
  Unknown | 1 | 0 | 1
Cancer Stage [Count of Participants; unit: Participants] — A diagnosis of advanced solid, incurable stage III or IV cancer was part of the eligibility criteria. Clinical staging without pathological confirmation of advanced disease was allowed. Cancer stage was collected on the "Tumor & Treatment Characteristics" measure which is completed at baseline by the clinical research associate under the direction of the oncology physician.
  Participants
    III | 28 | 19 | 47
    IV | 261 | 219 | 480
    Other | 3 | 10 | 13
    Unknown | 1 | 0 | 1
GA Impairments [Mean (Standard Deviation); unit: GA impairments] — There are 8 different GA domains in which impairments are measured, they include psychological status, cognition, social support, functional status, nutrition, co-morbidity, polypharmacy, and physical performance. The total number of GA-domain impairments were calculated. The total number of possible impairments range from 1-8 (patients had to have at least 1 GA impairment to be eligible for the study).
  GA impairments | 4.50 (1.54) | 4.45 (1.52) | 4.48 (1.53)
Number of Practice Sites [Number; unit: participants] | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Direct Communication About Age-related Concerns: Number of Discussions Related to the Geriatric Assessment That Occur in the Clinic Visit Between the Patient, Oncology Physician, and Caregiver. [Patient-Centered Outcomes Research Institute Specified]
Description: A geriatric assessment (GA), a validated set of patient-centered outcomes, has been shown to identify concerns (e.g., function, cognition) important to older persons with cancer and their caregivers. The geriatric assessment was used to define which age related topics discussed between patients and providers would be coded. We will apply linear mixed model methodology. The total number of conversations will be the response, and the arm will be the fixed effect. Estimation will be performed using Restricted Maximum Likelihood, and the null hypothesis of zero mean difference between arms will be tested using a F test. The specific NCORP practice site differences will be assessed graphically using Best Linear Unbiased Predictors (BLUP) of the mean response for each NCORP.
Time Frame: Baseline
Population: All baseline patients who were evaluable for this primary aim were included in this analysis.
  * Arm I patients excluded because 2 withdrew, 1 expired, 4 no audio captured and 2 primary aim protocol violations.
  * Arm II patients excluded (3 withdrew, 1 no audio captured).
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of Conversations
Groups:
- Arm I (GA Informational Intervention): Patients and their caregivers (if participating) complete the GA and receive the GA summary and recommendations guided by GA results provided by the oncology team to discuss and implement for each age-related issue at baseline.
  Informational Intervention:Complete GA summary plus GA-driven recommendations.
Arm/Group | Arm I (GA Informational Intervention) | Arm II (Usual Care)
Number analyzed (Participants) | 284 | 244
Number of Conversations | 8.02 [7.09 to 8.94] | 4.43 [3.42 to 5.44]
Statistical Analysis 1: Comparison: Arm I (GA Informational Intervention) vs Arm II (Usual Care); Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 3.59

2. Primary Outcome: Patient Satisfaction With Communication About Age-related Concerns: Measured by Health Care Climate Questionnaire (HCCQ). [NCI Specified]
Description: Will apply linear mixed model methodology. The total HCCQ scores will be the response, and the arm will be the fixed effect. HCCQ contains 7 questions, scale: 0-28. The higher the score the more satisfied the patients is with communication with their oncologists about age related concerns. Estimation will be performed using Restricted Maximum Likelihood, and the null hypothesis of zero mean difference between arms will be tested using a F test. The specific NCORP practice site differences will be assessed graphically using Best Linear Unbiased Predictors (BLUP) of the mean response for each NCORP.
Time Frame: Within 1-7 days of the baseline audio-recorded clinic consultation
Population: All baseline patients who were evaluable for this primary aim were included in this analysis.
  * Arm I patients excluded (2 patients withdrew, 19 patients with no HCCQ).
  * Arm II patients excluded (3 patients withdrew, 9 no HCCQ).
Measure: Least Squares Mean (95% Confidence Interval); unit: HCCQ total score
Arm/Group | Arm I (GA Informational Intervention) | Arm II (Usual Care)
Number analyzed (Participants) | 271 | 239
HCCQ total score | 23.34 [22.63 to 24.05] | 22.25 [21.49 to 23.01]
Statistical Analysis 1: Comparison: Arm I (GA Informational Intervention) vs Arm II (Usual Care); Test type: Superiority; p = 0.041, Mixed Models Analysis; Mean Difference (Final Values) = 1.09

3. Secondary Outcome: Geriatric Assessment (GA) Summary and GA Targeted-recommendations Provided to Patients, Caregivers and Oncology Physicians Prior to Their Treatment Influences Quality of Life of Older Patients Receiving Treatment and Their Caregivers.
Description: Patient Health Related Quality of Life (HRQoL) will be assessed with the Functional Assessment of Cancer Therapy-General (FACT-G) measured on a 0-108 scale with higher scores indicating a better outcome. We will apply linear mixed model methodology to compare the between arm differences.
Time Frame: Mean score over 4-6 weeks, 3 months, 6 months assessments following the intervention
Population: Enrolled patients who have completed the FACT-G
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I (GA Informational Intervention) | Arm II (Usual Care)
Number analyzed (Participants) | 286 | 241
units on a scale | 82.93 (0.71) | 83.16 (0.76)

4. Secondary Outcome: Geriatric Assessment (GA) Summary and GA Targeted-recommendations Provided to Patients, Caregivers and Oncology Physicians Prior to Their Treatment Influences Caregiver Satisfaction With Communication About Age-related Issues.
Description: We will compare the effect of the intervention on caregiver satisfaction (the modified health care climate questionnaire (HCCQ)- age for the caregiver, range 0-20; higher score better outcome). We will apply linear mixed model methodology to compare between arm differences.
Time Frame: At 4-6 weeks, 3 months and 6 months following the intervention
Population: The number of caregiver's with an available HCCQ at 4-6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Arm I (GA Informational Intervention) | Arm II (Usual Care)
Number analyzed (Participants) | 189 | 158
score on a scale
  4-6 Weeks | 16.44 (0.29) | 15.39 (0.31)
  3 months: number analyzed (Participants) | 166 | 139
  3 months | 16.47 (0.30) | 15.64 (0.32)
  6 months: number analyzed (Participants) | 150 | 111
  6 months | 16.49 (0.31) | 15.87 (0.34)
Statistical Analysis 1: Comparison: Arm I (GA Informational Intervention) vs Arm II (Usual Care); Test type: Superiority; p = 0.03, Mixed Models Analysis; The above p-values is for 4-6 weeks; Mean Difference (Final Values) = 1.05, 95% CI 2-sided [0.12 to 1.98] — The above values are for 4-6 weeks
Statistical Analysis 2: Comparison: Arm I (GA Informational Intervention) vs Arm II (Usual Care); Test type: Superiority; p = .08, Mixed Models Analysis; The above p-value is for is for 3 months; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [-0.11 to 1.77] — The above values are for 3 months
Statistical Analysis 3: Comparison: Arm I (GA Informational Intervention) vs Arm II (Usual Care); Test type: Superiority; p = 0.20, Mixed Models Analysis; The above p-value is for 6 months; Mean Difference (Final Values) = 0.62, 95% CI 2-sided [-0.36 to 1.59] — The above values are for 6 months

5. Secondary Outcome: Geriatric Assessment (GA) Summary and GA Targeted-recommendations Provided to Patients, Caregivers and Oncology Physicians Prior to Their Treatment Influences Quality of Life of Older Patients Receiving Treatment and Their Caregivers.
Description: Caregiver Health Related Quality of Life (burden) will be assessed with the Caregiver Reactions Assessment (CRA- [Overall scale ranges from 1-5, better or worse outcome depending on subscale- Self Esteem Subscale higher score indicates better outcome, Disrupted Schedule subscale lower score indicates better outcome, Financial problems subscale lower score indicates better outcome, Lack of Social Support subscale lower score indicates better outcome, Health Problems subscale lower score indicates better outcome]). We will apply linear mixed model methodology to compare between arm differences
Time Frame: Mean 4-6 weeks, 3 months, and 6 months after the intervention
Population: The number of caregivers with a CRA
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Arm I (GA Informational Intervention) | Arm II (Usual Care)
Number analyzed (Participants) | 229 | 182
units on a scale
  Self-Esteem | 4.41 (0.03) | 4.38 (0.03)
  Disrupted Schedule | 2.57 (0.05) | 2.58 (0.06)
  Financial Problems | 1.97 (0.04) | 2.04 (0.04)
  Lack of Social Support | 1.87 (0.04) | 1.91 (0.04)
  Health Problems | 1.98 (0.03) | 2.03 (0.04)

ADVERSE EVENTS:
Time Frame: Patients were followed for 6 months post-baseline during which time adverse events were collected.
Arm/Group | Arm I (GA Informational Intervention) | Arm II (Usual Care)
All-Cause Mortality (participants affected / at risk) | 42/296 | 30/250
Serious Adverse Events (participants affected / at risk) | 0/296 | 0/250
Other Adverse Events (participants affected / at risk) | 0/296 | 0/250

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT02107443/Prot_001.pdf
  • Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT02107443/SAP_000.pdf